CLINICAL TRIAL: NCT03122704
Title: Prevalence of Group B Streptococcus Infection in Pregnant Women Conceived Through IVF Diagnosed With Preterm Labor.
Brief Title: Group B Streptococcus (GBS) Infection and in Preterm Labor Women Conceived Through IVF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Manh Tuong Ho (Other)
Responsible Party: Sponsor-Investigator, Manh Tuong Ho, Doctor, Vietnam National University
Organization: Vietnam National University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NCKH/CGRH_09_2015
Record Dates: First submitted 2015-10-21; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Preterm Labor
MeSH Terms: conditions — Obstetric Labor, Premature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group B Streptococcus (GBS) screening (Experimental): Vaginal and anal swab of patients will be screened for GBS screening
  Interventions: Procedure: GBS screening

INTERVENTIONS:
Procedure: GBS screening — Vaginal and anal swabs of patients will be screened for GBS screening

SUMMARY:
This is a cross - sectional study to determine the prevalence of GBS infection and associated factors in preterm labor women conceived through ART.

221 subjects will be involved.

DETAILED DESCRIPTION:
Pregnant women at 20 0/7 to 36 6/7 weeks of gestation, conceived through ART, with signs and symptoms of preterm labor will be recruited.

Anal - vaginal fluid samples will be taken by 2 cotton swabs from each participant for culture. Digital examination will be performed after that. Only participants fulfilling all the study's eligible criteria will be interviewed face-to-face with a questionnaire.

The samples will be sent immediately to My Duc hospital laboratory or will be stored in Stuart-Amies medium in < 4 hours. All culture results are interpreted based on Clinical and Laboratory Standards Institute (CLSI) in 2012.

Statistical analysis was performed by Statistical Package for the Social Sciences (SPSS) v.20 and chi-square test. A p-value of < 0.05 was considered as statistically significant.

ELIGIBILITY:
* Inclusion Criteria:

To be eligible for enrolment into this trial, subject must fulfil all of the following criteria, unless specified otherwise

* Being conceived through IVF
* Moderate uterine contractions (2 contractions per 10 minutes, duration < 30 seconds)
* 20 0/7 to 36 6/7 weeks of gestation
* Intact membrane
* Cervical dilation ≤ 3 cm
* Willing to participate into the study

  * Exclusion Criteria:

To be eligible for enrolment in this study each subject must not meet any of the following criteria:

* Having had intercourse during 24 hours before
* Being suspected of amniotic leakage
* Rupture of membrane identified by direct observation through speculum examination of amniotic fluid flow from cervix
* Vaginal bleeding
* Being suspected of placenta abruption, placenta previa
* Having been treated with antibiotics within 1 week before
* Vaginal douche within 48 hours before
* Having used vaginal medicines during 48 hours before
* Having vaginal ultrasound shortly before
* Urine culture positive with GBS

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of women with GBS infection | 7 days after swab taken
  Number of women with GBS infection divided by total number of women under screening

CONTACTS AND LOCATIONS:
Overall Officials: Tuong M Ho, MD, Study Director — Research Center for Genetics and Reproductive Health
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Tan Binh District, Vietnam